CLINICAL TRIAL: NCT04768010
Title: Misoprostol for the Management of Bloating and Gaseous Distension in Patients With Cirrhosis: an Open Label Trial
Brief Title: Misoprostol for Bloating and Distension
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: After significant delays study was never initiated. No participants enrolled
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12715
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Distension; Gas Bloat Syndrome; Constipation
MeSH Terms: conditions — Dilatation, Pathologic; Gas bloat syndrome; Constipation | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Misoprostol (Experimental): Participants will receive 100-200 micrograms of oral misoprostol twice daily.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Participants will started by receiving 100 micrograms of oral misoprostol twice daily. If adverse effects are not noted dose can be titrated up to 200 micrograms of misoprostol twice daily. Participants will receive a total of five doses.
  Other Names: Cytotec (brand name)

SUMMARY:
Symptoms of bloating, abdominal distension, and constipation are common in patients with cirrhosis. These symptoms may be explained by disease-associated effects in gastrointestinal physiology, as well as medication side-effects. The presence of these symptoms affect quality of life, as well as risk for encephalopathy. Misoprostol is a synthetic prostaglandin approved for the treatment prevention of NSAID-induced gastric ulcers. The drug also causes smooth muscle contraction in the gastrointestinal tract has been shown to improve colonic motility.

This study aims to assess the efficacy of misoprostol for treating bloating, distension, and constipation in patients with cirrhosis. Study participants will receive misoprostol for a duration of three days. Participants will complete pre-intervention and post-intervention symptom questionnaires and low dose abdominal computed tomography (CT) scan. These measures will be used to assess subjective symptom scores and objective measurement of intestinal gas and colonic stool. Post-intervention measures will be compared to pre-intervention measures to assess improvement of symptoms.

DETAILED DESCRIPTION:
Specific Aims of Study:

To determine whether misoprostol is beneficial in patients with cirrhosis with bloating secondary to stool and gaseous distension, patient with marked symptoms that are refractory to standard of care will receive open label Misoprostol (100mcg twice daily and increased to 200mcg twice daily based on response) before and after 2 days of treatment with the following assessments:

1. Characterization of bloating and abdominal discomfort symptoms as assessed by the Patient Assessment of Constipation (PAC-SYM) and Patient Assessment of Gastrointestinal Symptoms (PAGI-SYM) Questionnaires composite scores and subscale scores before
2. Radiologic quantitation of intestinal gaseous distension as assessed by volumetric measurement of ultra-low radiation abdominal CT scan
3. Impact on severity of hepatic encephalopathy scores as assessed by West Haven criteria grading and Psychometric Hepatic Encephalopathy Score (PHES)

This study is a prospective, open-label trial comparing the efficacy of misoprostol in the management of bloating and gaseous distension in patients with cirrhosis.

The duration of the study will be over 3 days for each enrolled patient and will include an initial screening encounter prior to day 1 of the study period. During the screening encounter, participants' will receive a complete history and physical including review of treatment with standard of care treatments such as polyethylene glycol, bisacodyl, docusate, senna, and simethicone. If symptoms are not relieved by the use of these standard of care treatments participants will be fully screened, provided informed consent, enrolled in the trial.

Participants will be administered the PAC-SYM, PAGI-SYM questionnaires in addition to determination of West Haven Criteria Grade and PHES. These baseline demographics will be collected and used as reference for comparison of post-intervention questionnaire results. Baseline abdominal girth will also be documented. Afterwards, participants will receive a baseline low-dose abdominal CT for the volumetric assessment of intestinal gas. Abdominal X-ray available from CT data will be used for scoring of colonic stool burden.

Participants will be started on the study medication on day 1. On day 1, participants will receive an initial dose of 100 micrograms of misoprostol administered orally. The patient will be monitored for adverse effects and, if none observed, will continue 100 microgram dose twice daily with increase to 200mcg on day 2 if symptoms not improved. All primary outcomes will be assessed daily between morning and evening doses.

On the morning of day 3, participants will receive one dose of study drug at dose received on day 2. After administration of the drug, participants will repeat ultra-low dose abdominal CT and complete a final assessment with the PAC-SYM, PAGI-SYM, PHES and West Haven Grading.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Participants who voluntarily sign and date an informed consent
* Participants who are willing to adhere to the procedures in this protocol
* Have biopsy or strong clinical evidence for the presence of cirrhosis
* Report any of the following symptoms: abdominal bloating, distension, and/or constipation (<3 bowel movements per week)
* Have failed management with standard-of-care therapies used at Montefiore Medical Center
* Have received a standard-of-care abdominal x-ray revealing gaseous distension or fecal loading

Exclusion Criteria:

* hemodialysis
* active infection
* Evidence of bowel obstruction
* Evidence of moderate or large ascites
* history of bowel surgery, uncontrolled thyroid disorders, inflammatory bowel disease
* pregnancy
* intubation during current hospitalization
* inability to provide informed consent.
* History of allergic reaction to prostaglandins
* Patients on narcotic medications besides a stable dose of methadone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Change in Patient Assessment of Gastrointestinal Symptoms (PAGI-SYM) Questionnaire Score | Baseline, Day 2, and Day 3
  The PAGI-SYM is a validated 20 item self-report questionnaire divided in to six domains: heartburn/regurgitation, fullness/early satiety, nausea/vomiting, bloating, upper abdominal pain, and lower abdominal pain. Scores for each question range from 0 (none absent) to 5 (very severe). This questionnaire obtains subscale scores derived from the average scores across these six domains. The original questionnaires asks "How severe have each of these following symptoms been in the past two weeks?" For the purpose of this study, we have obtained manufacturer approval to modify the questionnaire to ask about symptoms severity in the past day.
Change in Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire Score | Baseline, Day 1, Day 2, and Day 3
  The PAC-SYM is a validated 12 item self-report questionnaire divided into abdominal, rectal, and stool domains. The questionnaire has 4 items for abdominal symptoms, 3 items for rectal symptoms, and 5 items for stool symptoms. Scores range from 0 (none or absent) to 4 (very severe). The total score is the mean of the individual item scores.The original questionnaires asks "How severe have each of these following symptoms been in the past two weeks?" For the purpose of this study, we have obtained manufacturer approval to modify the questionnaire to ask about symptoms severity in the past day.

SECONDARY OUTCOMES:
Change in intestinal gas volume from baseline to post-intervention | Baseline and Day 3
  Measured by low dose abdominal CT
Change in stool burden from baseline to post-intervention | Baseline and Day 3
  Scored using abdominal X-ray
Change in Abdominal Girth | Baseline, Day 1, Day 2, and Day 3
  Abdominal girth will be measured in centimeters using a tape measure.
Change in Psychometric Hepatic Encephalopathy Score (PHES) | Baseline, Day 2, and Day 3
  The PHES is a series of five neuropsychological tests used in the diagnosis of minimal hepatic encephalopathy. The tests used in this score include the digit-symbol test, number connection tests A and B, the serial dotting test, and the line-drawing test. The final score for the PHES is derived from the sum of the scores of these individual tests. To determine individual test scores, the difference between the predicted and observed results for each test are divided by the corresponding standard deviation (SD) for the reference population to obtain the deviation from 'normal' as a multiple of the SD. Final scores range from -15 to +5. Lower scores are found in patients with encephalopathy, with a score <-4 SD being considered to represent the presence of minimal hepatic encephalopathy.
Change in Abdominal Pain | Baseline, Day 2, and Day 3
  The severity of abdominal pain will de determined from the individual Likert score derived from the Patient Assessment of Gastrointestinal Symptoms (PAGI-SYM). The Likert scale ranges from Scores for each question range from 0 (none absent) to 5 (very severe).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No